CLINICAL TRIAL: NCT03939832
Title: Effect of Intraoperative Oxygen Tension on Patient Outcomes After Cardiac Surgery With Cardiopulmonary Bypass: a Pilot Study
Brief Title: FiO2 and Outcomes After Cardiac Surgery With Cardiopulmonary Bypass
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 pandemic, it was no possible to recruit patients for this study.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor of Anesthesiology and Pain Medicine, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FiO2 CPB
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Patients Undergoing Cardiac Surgery Using Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FiO2 0.5 (Active Comparator)
  Interventions: Other: Fraction of inspired oxygen level
- FiO2 1.0 (Active Comparator)
  Interventions: Other: Fraction of inspired oxygen level

INTERVENTIONS:
Other: Fraction of inspired oxygen level — A fraction of inspired oxygen level during cardiac surgery using cardiopulmonary bypass will be set differently: 0.5 versus 1.0.

SUMMARY:
Conventionally, a relatively high level of fraction of inspired oxygen (FiO2) has been used for secure a margin of safety in patients undergoing cardiac surgery using cardiopulmonary bypass (CPB). Since the potential adverse effects of hyperoxemia (via reactive oxygen species, vasocontriction, perfusion heterogeneity, myocardiac injury, etc.), various studies on this topic has been performed. However, the results are conflicting and inconsistent, and the consensus about whether the use of additional oxygen supply in cardiac surgery using CPB has not been reached among practitioners yet.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for cardiac surgery using cardiopulmonary bypass

Exclusion Criteria:

* Planned implementation of deep hypothermic circulatory arrest
* Preoperative respiratory support with the fraction of inspired oxygen of 0.5 and more.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
hospital LOS | From the beginning of surgery until the hospital discharge after surgery through study completion, an expected average of two weeks
  length of hospital stay after cardiac surgery using cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea